CLINICAL TRIAL: NCT07392658
Title: Phase II Trial of Amivantamab Plus Monochemotherapy in Platinum Unfit NSCLC Patients With EGFR exon20 Insertion Mutations.
Acronym: AMICUTE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMICUTE
Record Dates: First submitted 2025-11-24; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Metastatic NSCLC - Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab

STUDY DESIGN:
Intervention Model Description: This is a phase II multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMIVANTAMAB (Experimental)
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Amivantamab — Subcutaneous amivantamab at the dose of 1600 mg (2240 mg, ≥80 kg) on cycle 1 day 1, than at the dose of 2400 mg (3360 mg, ≥80 kg) on cycle 1 day 8 and 15 and than every 3 weeks starting from cycle 2 day 1, in combination with monochemoterapy (investigator's choice between pemetrexed 500 mg/m2 IV Q3W or gemcitabine 1000 mg/m2 IV day 1-8 Q3W)

SUMMARY:
To assess safety and efficacy of amivantamab plus monochemotherapy in terms of ORR, PFS and OS in subjects with EGFR exon20 insertion mutations metastatic non-small cell lung cancer unfit for platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is a phase II multicenter study assessing efficacy and safety of amivantamab plus monochemotherapy in patients with EGFR exon20 insertion mutations metastatic NSCLC who are unfit for platinum-based chemotherapy. After evaluation of all inclusion and exclusion criteria and after informed consent signature all eligible patients will be treated with subcutaneous amivantamab at the dose of 1600 mg (2240 mg, ≥80 kg) on cycle 1 day 1, than at the dose of 2400 mg (3360 mg, ≥80 kg) on cycle 1 day 8 and 15 and than every 3 weeks starting from cycle 2 day 1 in combination with monochemoterapy (investigator's choice between pemetrexed or gemcitabine), until disease progression, unacceptable toxicity or patient refusal. Disease assessment will be performed every 8 weeks. Response will be evaluated according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Male or female patient aged ≥18 years;
* Histologically or cytologically confirmed stage IV or recurrent non-squamous NSCLC harboring EGFR exon20 insertion mutation;
* No prior systemic treatment;
* Unfit for platinum-based chemotherapy; Unfit for platinum is defined by a glomerular filtration rate (GFR) value less than 50 ml/min/BSA (body surface area) 1.73 m2 (or a CCR value of <50 ml/min) or age 80 years, presence of neurological disorders or hypersensitivity to platinum.
* At least one radiological measurable disease according to RECIST criteria version 1.1;
* Patients with brain metastases are eligible if they are asymptomatic and stable (i.e. without evidence of progression by imaging for at least two weeks prior to the first dose of trial treatment and without deterioration of any neurologic symptoms);
* Performance status 0-2 (ECOG PS);
* Patient compliance to trial procedures;
* Adequate bone marrow function (ANC ≥ 1.5x109/L, platelets ≥75x109/L, haemoglobin >9 g/dl);
* Adequate liver function (Total bilirubin ≤1.5 x ULN; subjects with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits, transaminases no more than 3xULN/<5xULN in presence of liver metastases);
* Normal level of alkaline phosphatase and Serum creatinine <1.5 x ULN and creatinine clearance >45 mL/min as measured or calculated; refer to Appendix --Cockcroft-Gault Formula for Estimated creatinine clearance 12 Patients should be using adequate contraceptive measures, should not be breastfeeding, until 7 months after the last dose, and must have a negative pregnancy test (serum or urine) prior to first dose of study drug (within 72 hours) and must agree to further serum or urine pregnancy tests during the study; or female patients must have an evidence of non-childbearing potential by fulfilling one of the following criteria at screening: Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments; Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution.

A participant must be either of the following:

* Not of childbearing potential
* Of child-bearing potential and practicing true abstinence during the entire period of the study, including up to 6 months after the last dose of study treatment is given
* Of childbearing potential and practicing 2 methods of contraception, including 1 highly effective user independent method and a second method (examples of highly effective methods of contraception are in section 9.6: Contraceptive Guidance and Collection of Pregnancy Information).

A participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study treatment.

A participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for 6 months after receiving the last dose of study treatment. A participant who is sexually active with a partner of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and their partner must also be practicing a highly effective method of contraception (ie, established use of oral, injected, or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]).

If the participant is vasectomized, they must still use a condom (with or without spermicide) for prevention of passage of exposure through ejaculation, but their partner is not required to use contraception.

A participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study treatment.

Note: If the childbearing potential changes after start of the study (eg, participant of childbearing potential who is not heterosexually active becomes active, premenarchal participant experiences menarche) the participant must begin birth control, as described above.

Exclusion Criteria:

* Uncontrolled infectious liver disease;
* Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg) Note: participants with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.
* Positive hepatitis C antibody (anti-HCV). Note: participants with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
* Participant is positive for human immunodeficiency virus (HIV), with 1 or more of the following:

Receiving ART that may interfere with study treatment (consult sponsor for review of medication prior to enrollment) CD4 count <350 at screening AIDS-defining opportunistic infection within 6 months of start of screening Not agreeing to start ART and be on ART>4 weeks plus having HIV viral load <400 copies/mL at end of 4-week period (to ensure ART is tolerated and HIV controlled).

-Participant has active cardiovascular disease including, but not limited to: A medical history of deep vein thrombosis or pulmonary embolism within 1 month prior to randomization or any of the following within 6 months prior to randomization: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome. Clinically non-significant thrombosis, such as non-obstructive catheter-associated thrombus, incidental or asymptomatic pulmonary embolism, are not exclusionary.

* Uncontrolled (persistent) hypertension: systolic blood pressure >160 mm Hg; diastolic blood pressure >100 mm Hg.
* Congestive heart failure (CHF), defined as New York Heart Association (NYHA) class III-IV or hospitalization for CHF (any NYHA class; refer to Appendix 6: New York Heart Association Criteria) within 6 months of randomization.
* Participant has an uncontrolled illness, including but not limited to:

Uncontrolled diabetes Ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to starting study treatment] or diagnosed or suspected viral infection.

Active bleeding diathesis Impaired oxygenation requiring continuous oxygen supplementation Psychiatric illness, social situation, or any other circumstances that would limit compliance with study requirements Any ophthalmologic condition that is clinically unstable

* Absence of measurable lesions;
* Concomitant radiotherapy;
* Previous treatment with any EGFR Exon20ins-targeted TKIs;
* Symptomatic or immediately requiring therapy for brain metastases or carcinomatous meningitis. Subjects with asymptomatic and stable or treated brain metastases may participate;
* Participant has concurrent or prior malignancy other than the disease under study. The following exceptions require consultation with the Medical Monitor:

  1. Non-muscle invasive bladder cancer (NMIBC) treated within the last 24 months that is considered completely cured.
  2. Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured.
  3. Non-invasive cervical cancer treated within the last 24 months that is considered completely cured.
* Participant had major surgery excluding placement of vascular access or tumor biopsy, or had significant traumatic injury within 4 weeks before randomization, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study.

Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate.

* History of extensive disseminated/bilateral or known presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis;
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV);
* Pregnancy or lactating female;
* Other serious illness or medical condition potentially interfering with the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
ORR | "through study completion, an average of 1 year"
  Objective Response Rate (ORR) according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- I.F.O. Istituti Fisioterapici Ospitalieri Istituto Nazionale Tumori "Regina Elena", Medical Oncology 2, Roma, Roma (RM), Italy